CLINICAL TRIAL: NCT02420951
Title: Local Injection of Local Anesthetic 24 Hours After Knee Replacement Surgery
Brief Title: Local Injection of Local Anesthetic 24 Hours After Knee Replacement Surgery May Decrease Pain for Several More Hours
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Wolfgang Fitz, Associate Orthopedic Surgeon, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Injection after total knee
Record Dates: First submitted 2015-01-28; First posted 2015-04-20 (Estimated); Results first posted 2017-03-31 (Actual); Last update posted 2018-01-12 (Actual); Status verified 2017-12

CONDITIONS: Arthroplasty, Knee; Pain
Keywords: Knee; Arthroplasty; Bupivacaine; Anesthetics, Local
MeSH Terms: conditions — Pain | interventions — Bupivacaine

STUDY DESIGN:
Intervention Model Description: We randomized 50 patients undergoing TKA at one institution into two groups. Group 1, 25 patients, received a postoperative intra-articular catheter in combination with injection of 30 ml of 0.5% Marcaine the day after surgery before removal. Group 2, 25 patients, received no pain catheter. Both groups received intraoperative pericapsular injection and postoperative pain medication. We measured pain scores using the Visual Analog Scale (VAS) and recorded narcotic medication consumption in morphine milligram equivalents (mgs).
Oversight: Data Monitoring Committee: No

ARMS (2):
- Injection (Experimental): Will receive injection of 30ml of .5% bupivacaine solution prior to catheter removal
  Interventions: Drug: Bupivacaine
- No Injection (Active Comparator): Will not receive injection of bupivacaine prior to catheter removal
  Interventions: Other: No Intervention

INTERVENTIONS:
Drug: Bupivacaine — Injection of local anesthetic immediately prior to catheter removal, 24 hours postop.
  Other Names: marcaine
  Arms: Injection
Other: No Intervention — No injection of local anesthetic immediately prior to catheter removal, 24 hours postop.
  Arms: No Injection

SUMMARY:
The purpose of this study is to determine if an additional injection of local anesthetic immediately prior to removal of the local anesthetic infiltration catheter on postoperative day one is effective in increasing pain reduction, patient satisfaction or outcome measures following total knee replacement (TKR). It is hypothesized that an additional injection of 30ml of .5% bupivacaine solution immediately before infiltration catheter removal will provide pain reduction, patient satisfaction and outcome measures equal or superior to catheter removal with no additional injection.

Patients who are undergoing unilateral total knee replacement (TKR) and choose to participate will be randomly assigned to a treatment group.Patients in group one (treatment group) will receive a 30ml dose of .5% bupivacaine solution injected into the local anesthetic infiltration catheter immediately prior to its removal on postoperative day one. Patients in group two (control group) will receive no additional medication during local anesthetic infiltration catheter removal.

DETAILED DESCRIPTION:
The purpose of this study is to determine if an additional injection of local anesthetic immediately prior to removal of the local anesthetic infiltration catheter on postoperative day one is effective in increasing pain reduction, patient satisfaction or outcome measures following total knee replacement (TKR). It is hypothesized that an additional injection of 30ml of .5% bupivacaine solution immediately before infiltration catheter removal will provide pain reduction, patient satisfaction and outcome measures equal or superior to catheter removal with no additional injection. The target enrollment for this study is 50 participants, 25 in each of groups one and two.

Patients who are undergoing unilateral total knee replacement (TKR) at Brigham and Women's Faulkner Hospital and meet all eligibility criteria will be informed about the study and asked if they would like to participate. Upon agreement, patient's consent will be obtained and they will be randomly assigned to a treatment group. Patients in group one (treatment group) will receive a 30ml dose of 0.5% bupivacaine solution injected into the local anesthetic infiltration catheter immediately prior to its removal on postoperative day one. Patients in group two (control group) will receive no additional medication during local anesthetic infiltration catheter removal.

Members of both groups will be asked to complete Visual Analog Scale (VAS) pain and satisfaction surveys and also to track daily narcotic pain medication consumption during the first week postoperatively. Measures of swelling in the operative knee will be collected for members of both groups at the first routine postoperative appointment approximately one week after surgery. Swelling will be measured using a Perometer which calculates the total volume of the extremity in cubic centimeters (Pero-System, Wuppertal, Germany). Proprioception will be measured using a SD Balancer (Biodex Medical Systems, Shirley, NY) which calculates the the overall stability index (OSI) and compares it to age standardized data. Quadriceps strength using a handheld dynamometer. Outcome measures will be collected for members of both groups prior to surgery and at the second routine postoperative appointment between 6 weeks after surgery. Swelling will be also measured at the first post-operative visit 1 week after surgery. These data measures, as well as any complications will be recorded and used for analysis at the completion of the study.

The Principal Investigator (PI) will review all pain, satisfaction, narcotic usage and proprioception data on a weekly basis with the research assistant (RA) as it is collected. These checks will help to ensure validity and patient safety. Privacy and confidentially will be assured by using codes as deidentifiers in place of identifying information on any data sheets used in analysis. Data which identifies the patient will be made available only to investigators and stored only in a private folder on department computers protected with a firewall. No data will be shared outside of Partners. Adverse events will be promptly reported to the PHRC as per PHRC rules.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Undergoing unilateral knee replacement
* If female, not pregnant
* Agree to participate in the follow-up appointment
* Understand and sign the informed consent form

Exclusion Criteria:

• Bilateral TKA planned

* Use of narcotic medication before surgery
* Any other surgery within the three months prior to TKR
* Inflammatory arthritis
* Any chronic pain conditions or problems, including but not limited to chronic back pain, fibromyalgia or multiple sclerosis
* Osteoarthritis of the non-operative knee
* Osteoarthritis of one or both hips

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-10-05 (Actual); Primary Completion 2016-03-22 (Actual); Study Completion 2016-12-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Fitz, MD, Principal Investigator — Brigham and Women's Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chaumeron A, Audy D, Drolet P, Lavigne M, Vendittoli PA. Periarticular injection in knee arthroplasty improves quadriceps function. Clin Orthop Relat Res. 2013 Jul;471(7):2284-95. doi: 10.1007/s11999-013-2928-4. Epub 2013 Mar 21. PMID 23516031
- [Background] Barrington JW, Halaszynski TM, Sinatra RS, Expert Working Group On Anesthesia And Orthopaedics Critical Issues In Hip And Knee Replacement Arthroplasty FT. Perioperative pain management in hip and knee replacement surgery. Am J Orthop (Belle Mead NJ). 2014 Apr;43(4 Suppl):S1-S16. PMID 24911869
- [Background] Teng Y, Jiang J, Chen S, Zhao L, Cui Z, Khan MS, Du W, Gao X, Wang J, Xia Y. Periarticular multimodal drug injection in total knee arthroplasty. Knee Surg Sports Traumatol Arthrosc. 2014 Aug;22(8):1949-57. doi: 10.1007/s00167-013-2566-0. Epub 2013 Jun 20. PMID 23783531
- [Background] Jiang J, Teng Y, Fan Z, Khan MS, Cui Z, Xia Y. The efficacy of periarticular multimodal drug injection for postoperative pain management in total knee or hip arthroplasty. J Arthroplasty. 2013 Dec;28(10):1882-7. doi: 10.1016/j.arth.2013.06.031. Epub 2013 Aug 1. PMID 23910819
- [Background] National Center for Health Statistics. National Hospital Discharge Survey, 2010. Hyattsville, Maryland: Public Health Service. 2010.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Injection | No Injection
Started | 25 | 25
Completed | 25 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Injection | No Injection | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 9 | 16
  >=65 years | 18 | 16 | 34
Age, Continuous [Mean (Full Range); unit: years] | 68.96 [57 to 81] | 66.44 [50 to 79] | 67.7 [50 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 14 | 29
  Male | 10 | 11 | 21

OUTCOME MEASURES:

1. Primary Outcome: Pain Assessed Using the VAS 0-10 Pain Scale
Description: Pain will be assessed using the VAS 0-10 pain scale. 0 is no pain and 10 in worst imaginable pain.
Time Frame: 7 days
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Injection | No Injection
Number analyzed (Participants) | 25 | 25
units on a scale | 2.763 [1.99 to 3.33] | 2.483 [1.89 to 2.89]

2. Secondary Outcome: Pain Med Consumption Assessed Using Questionnaire/Hospital Records
Description: Questionnaire/Hospital Records - While patients are in the hospital, pain medication consumption will be tracked in their electronic medical record. At home, patients will be asked to keep a log of pain medication consumption. They will be asked to record this information on a questionnaire at their first post-operative visit.
Time Frame: 2 days
Measure: Mean (Full Range); unit: morphine milligram equivalents (mgs)
Arm/Group | Injection | No Injection
Number analyzed (Participants) | 25 | 25
morphine milligram equivalents (mgs) | 79.45548 [9.0 to 185.64] | 62.39041 [5.0 to 212.5]

3. Secondary Outcome: Pain Med Consumption Assessed Using Questionnaire/Hospital Records
Description: Total pain medications consumed by the patient, determined through the patients' own records in the questionnaire as well as hospital records of pain med administration and prescription.
Time Frame: 7 days
Population: Data were not collected.
Arm/Group | Injection | No Injection
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Swelling Measured Using a Perometer
Description: Swelling in the affected TKR joint, as measured by a perometer.
Time Frame: 7 days
Population: Data were not collected.
Arm/Group | Injection | No Injection
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Proprioception Measured Using a SD Balancer
Description: Proprioception measured after surgery, as measured by an SD balancer.
Time Frame: 7 days
Population: Data were not collected.
Arm/Group | Injection | No Injection
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Quadriceps Strength Measured Using a Biodex Handheld Dynamometer"
Description: Quadriceps strength after surgery, as measured by a Biodex handheld dynamometer.
Time Frame: 7 days
Population: Data were not collected.
Arm/Group | Injection | No Injection
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Injection | No Injection
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No